CLINICAL TRIAL: NCT00780507
Title: Fecal Biomarker Study for Patients From a Once Daily Study for Efficacy in a Ulcerative Colitis Maintenance Study
Brief Title: Fecal Biomarker Study for Patients With Ulcerative Colitis
Status: Completed | Type: Observational
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Other Study IDs: 2007096
Record Dates: First submitted 2008-10-24; First posted 2008-10-27 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Human feces protein biomarkers Enrollment is number of specimens rather than number of subjects
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients are in a state of remission
- 2: Patients are in a flare

SUMMARY:
The present study will analyze fecal levels of FC and FL in UC patients who relapse (flare) while on a QD or a BID Asacol treatment regimen and compare those levels to levels of FC and FL in UC patients who do not relapse (flare).

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for this biomarker study;
* Be enrolled in Study 2007021 (QDIEM).

Exclusion Criteria:

* Meet the QDIEM Protocol 2007021 for Exclusion Criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of ulcerative colitis patients willcome from clients within the United States and are participants in the QDIEM Asacol study (2007021/NCT00505778)
Sampling Method: Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2007-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Compare the fecal biomarker calprotectin between the UC patients who relapse (flare) and the UC patients who remain in remission throughout the study while on Asacol regardless of the maintenance regimen. | one year

SECONDARY OUTCOMES:
To compare the fecal levels of the 2 biomarkers (FC and FL) in patients who are on BID and QD treatment regimens and who remain in remission for the duration of the study; | one year

CONTACTS AND LOCATIONS:
Overall Officials: William S Aronstein, MD, PhD, Study Director — Procter and Gamble
Locations (59):
- United States (59):
  - Research Facility, Lowell, Arkansas
  - Research Facility, Anaheim, California
  - Research Facility, Folsom, California
  - Research Facility, Los Angeles, California
  - Research Facility, Merced, California
  - Research Facility, San Diego, California
  - Research Facility, Upland, California
  - Research Facility, Lafayette, Colorado
  - Research Facility, Torrington, Connecticut
  - Research Facility, Fort Lauderdale, Florida
  - Research Facility, New Port Richey, Florida
  - Research Facility, Palm Harbor, Florida
  - Research Facility, Tampa, Florida
  - Research Facility, Zephyrhills, Florida
  - Research Facility, Decatur, Georgia
  - Research Facility, Marietta, Georgia
  - Research Facility, Newnan, Georgia
  - Research Facility, Arlington Heights, Illinois
  - Research Facility, Oak Lawn, Illinois
  - Research Facility, Urbana, Illinois
  - Research Facility, South Bend, Indiana
  - Research Facility, Clive, Iowa
  - Research Facility, Topeka, Kansas
  - Research Facility, Bowling Green, Kentucky
  - Research Facility, Shreveport, Louisiana
  - Research Facility, Lutherville, Maryland
  - Research Facility, Braintree, Massachusetts
  - Research Facility, Chesterfield, Michigan
  - Research Facility, Rochester Hills, Michigan
  - Research Facility, Jefferson City, Missouri
  - Research Facility, Egg Harbor, New Jersey
  - Research Facility, Babylon, New York
  - Research Facility, Binghamton, New York
  - Research Facility, Cheektowaga, New York
  - Research Facility, Forest Hills, New York
  - Research Facility, Lake Success, New York
  - Research Facility, Pittsford, New York
  - Research Facility, Port Jefferson Station, New York
  - Research Facility, Boone, North Carolina
  - Research Facility, Morganton, North Carolina
  - Research Facility, New Bern, North Carolina
  - Research Facility, Raleigh, North Carolina
  - Research Facility, Canton, Ohio
  - Research Facility, Cincinnati, Ohio
  - Research Facility, Indiana, Pennsylvania
  - Research Facility, Lancaster, Pennsylvania
  - Research Facility, Warwick, Rhode Island
  - Research Facility, Jackson, Tennessee
  - Research Facility, Greenville, Texas
  - Research Facility, Houston, Texas
  - Research Facility, Lewisville, Texas
  - Research Facility, Longview, Texas
  - Research Facility, Odessa, Texas
  - Research Facility, Pasadena, Texas
  - Research Facility, Plano, Texas
  - Research Facility, Alexandria, Virginia
  - Research Facility, Chesapeake, Virginia
  - Research Facility, Winchester, Virginia
  - Research Facility, Spokane, Washington